CLINICAL TRIAL: NCT04803552
Title: Identification of Patients With Clinically Relevant Sleep Apnea With a Contactless Device in Rehabilitation Clinic
Brief Title: Non-contact Sleep Apnea Identification in Neurological Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sleepiz AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20-025-EX-KSM Bad Zurzach
Record Dates: First submitted 2021-03-16; First posted 2021-03-17 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Sleep Apnea; Stroke
Keywords: stroke; sleep apnea; contactless; screening
MeSH Terms: conditions — Sleep Apnea Syndromes; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contactless sleep apnea screening vs respiratory polygraphy (Experimental)
  Interventions: Device: Overnight sleep study with Sleepiz One and a respiratory polygraphy

INTERVENTIONS:
Device: Overnight sleep study with Sleepiz One and a respiratory polygraphy — Participants will undergo a screening night with Sleepiz One. and with a cardiorespiratory polygraphy device (Miniscreen, Heinen-Löwenstein).
  Measurements (Miniscreen, Heinen-Löwenstein)
  * Thoracic respiratory effort: respiration frequency (BR), respiration curve
  * Airflow: respiration frequency (BR), respiration curve
  * Body movement: body position
  * Blood oxygen saturation (SpO2)
  * Pulse
  Measurements (Sleepiz One):
  • Movement originating from breathing and heart contractions

SUMMARY:
To improve the quality of medical care in the group of poststroke patients, we are planning to examine neurological patients in a rehabilitation clinic simultaneously with a non-contact method (Sleepiz One) and a standard diagnostic polygraphy measurement. This easy and comfortable pre-screening (Sleepiz One) should reduce the barrier for ward physicians to request a sleep study. The method could help to overcome the bottleneck of resource-intense procedures. It is simple to carry out and does not disturb the sleep of the patients.

The scoring is done according to the AASM Manual Version 2.6. Patients with a confirmed diagnosis will be informed about therapy options by a sleep physician and receive a recommendation for further therapy in the discharge letter from the rehabilitation clinic.

The goal of the study is then to evaluate if a non-contact method, the Sleepiz One, presents an opportunity for a fast and easy pre-screening during rehabilitation. Therefore, the precision of binary classification of subjects based on their sleep apnea severity (AHI >= 15) made by Sleepiz One will be compared to PG data manually scored by expert sleep scorers.

ELIGIBILITY:
Inclusion Criteria:

* Age >18years
* Ability and consent to undergo electrophysiological routine assessment
* Informed Consent as documented by signature
* In-patients of RehaClinic Bad Zurzach

Exclusion Criteria:

* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Cardiac pacemaker or another implanted electrical device
* Women who are pregnant or breastfeeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, delirium etc. of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Binary classification of the apnea severity | 1 night
  Precision of binary classification of subjects based on their sleep apnea severity (apnea-hypopnea index (AHI) >= 15) made by Sleepiz One, compared to PG data manually scored by expert sleep scorers

CONTACTS AND LOCATIONS:
Overall Officials: Jens Acker, Dr., Principal Investigator — KSM Bad Zurzach
Locations (1):
- KSM Bad Zurzach, Bad Zurzach, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No